CLINICAL TRIAL: NCT06079710
Title: Jiangxi Provincial Children's Hospital
Brief Title: Effect of Intraoperative and Awakening Electroencephalogram on Awakening Agitation After General Anesthesia in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Other Study IDs: 2023-EEG-children
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Emergence Agitation; Anesthesia; Children's Surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergence agitation group
- Non emergence agitation group

SUMMARY:
The purpose of this study was to analyze the relationship between intraoperative and awakening electroencephalogram waveforms and awakening agitation after general anesthesia in children

ELIGIBILITY:
Inclusion Criteria:

1. The age of the child is 1-10 years old, regardless of gender;
2. ASA grading I to II;
3. Children undergoing hernia, appendix, or small orthopedic surgery under selective general anesthesia

Exclusion Criteria:

1. Respiratory infection occurred within 1 week before surgery;
2. Potential or existing contraindications to general anesthesia;
3. Significant abnormalities in blood routine or biochemical indicators;
4. Patients with cognitive function, mental illness, or neurodevelopmental delay;
5. Unable to cooperate in completing the test, the child's guardian refused to participate;
6. Other reasons why researchers believe it is not suitable to participate in this experiment.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who meet the inclusion criteria for surgery at Jiangxi Provincial Children's Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence agitation | The entire period from entering the recovery room to leaving the recovery room. Approximately 10 min-2 hours
  The level of postoperative emergence agitation (EA) was assessed using the pediatric anesthesia emergence delirium Scale (PAED) and the emergence agitation 5 Scale immediately after extubation, and then every 15 min until the child was returned to the ward.
  emergence agitation was defined as a PAED score of ≥12 or a emergence agitation 5 scale of >3.

SECONDARY OUTCOMES:
emergence time | Approximately 5 min-2 hours
  The period of time between the cessation of the use of anesthetic drugs and the recovery of the child's autonomous consciousness and the ability to respond correctly to external stimuli.
Postoperative pain intensity | The entire period from entering the recovery room to leaving the recovery room. Approximately 10 min-2 hours
  Immediately after postoperative recovery, assess the pain intensity of the child using the FLACC pain scale, and then evaluate again every 15 minutes until the child leaves the recovery room. FLACC is divided into 0-10 points
Compatibility during anesthesia induction period | Anesthesia induction period, up to 2 minutes
  The degree of cooperation between the patient and the doctor's instructions during anesthesia induction period. Using the Anesthesia Induction Cooperation Scale (ICC) for evaluation, the higher the ICC score, the worse the compatibility

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi Provincial, China